CLINICAL TRIAL: NCT00263705
Title: Adjuvant Capecitabine in Elderly Patients With Breast Cancer: a Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Chantal Bernard, Institut Jules Bordet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Elderly capecitabine 1
Record Dates: First submitted 2005-09-13; First posted 2005-12-09 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Elderly Patients; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capecitabine (Experimental): capecitabine 2000 mg/m² daily
  Interventions: Drug: Adjuvant capecitabine; Drug: capecitabine in aduvant setting

INTERVENTIONS:
Drug: Adjuvant capecitabine — Capecitabine 2000 mg/m² daily six cycles
  Other Names: Xeloda
Drug: capecitabine in aduvant setting — capecitabine in aduvant setting in ederly with breast cancer
  Other Names: Xeloda

SUMMARY:
Determination of guidelines regarding the use of adjuvant chemotherapy for early breast cancer in this population of Patients over 70 years old.

DETAILED DESCRIPTION:
Patients over 70 years old are under represented in clinical trials and there are no clear guidelines regarding the use of adjuvant chemotherapy for early breast cancer in this population. Whether CT retains the benefit conferred to younger patients remains uncertain. Moreover, there is extensive data regarding the increasing incidence and severity of side effects, such as myelotoxicity, mucositis and cardiotoxicity, with CT in this population. The efficacy and safety of CT in aged patients have been evaluated in different studies, most of them in haematological malignancy. Clearly, the patients' functional declines with age and the risk for CT toxicity rises with age. There is no standard of care regarding adjuvant chemotherapy for breast cancer in patients older than 70 years old.

This is a pilot study evaluating the feasibility and safety of 6 cycles of capecitabine in patients aged 70 years or more with high-risk early invasive breast cancer who have undergone optimal surgery.

The primary end point is to evaluate the possibility of delivering 6 cycles of capecitabine at the dose of 1000 mg/m² BID days 1 to 14 every 3 weeks, in terms of rate of patients who will receive an acceptable relative dose intensity (RDI).

Secondary end points are safety (including the evaluation of possible impact of treatment on the functional, cognitive and emotional status of the patient) and evaluating if some form of geriatric assessment add any information to the classic "inclusion criteria screening" in terms of prediction of treatment compliance and toxicity.

The study is being conducted at the Jules Bordet Institute. The planned accrual is 43 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ³70 years
2. Histologic diagnosis of early breast cancer for which the treating physician considers adjuvant chemotherapy to be beneficial. Recommended situations are for example:

   * endocrine non responsive (ER- and PgR -) and pT>1 cm, any T if N+ OR
   * endocrine responsiveness doubtful (ER and/or PgR- or poor [3 to-5 according to Harvey score (12) or £ 30% of positive cells by immunohistochemistry) and other risk factors (pT³2 cm or N+ or G3 or Her-2/neu positive, etc.) OR
   * endocrine responsive (ER and PgR > 5 according to Harvey score or > 30% of positive cells by immunohistochemistry) and at least two risk factors (pT³ 2 cm, N+, G3, Her-2/neu positive, etc.) OR
   * Very high risk (N>3) any ER/PgR.
3. ECOG Performance status £ 1
4. No previous exposition to chemotherapy in the neoadjuvant setting
5. Adequate organ function including:

   1. neutrophils ³ 1.5 x 109 /l
   2. platelets ³100 x 109 / l
   3. bilirubin < 1.25 x upper normal limit for the institution
   4. transaminases < 2.5 x upper normal limit for the institution
   5. calculated creatinine clearance of > 30ml/min (using the Crockoft and Gault formula)
   6. absence of

      * symptomatic ventricular arrhythmias;
      * clinically significant Congestive Heart Failure;
      * clinical and/or ECG evidence of myocardial infarction within the last 12 months;
      * Coronary artery disease requiring medication.
6. Absence of any psychological, familial or sociological condition or comorbidities that may affect compliance
7. Written informed consent obtained according to local ethics committee guidelines -

Exclusion Criteria:

N/A-

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
safety of capecitabine in ederly | 1 year
  safety of capecitabine in ederly

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Bernard, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium